CLINICAL TRIAL: NCT07335354
Title: Breast Reconstruction Decision Aid (RECONJOINT)
Brief Title: A Study of a Decision Tool for People Considering Breast Reconstruction Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25-079
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Focus Group Participants (No Intervention): Participants will receive usual care
- RECONJOINT/RCT Participants (Patients) (Experimental): Participants in the RECONJOINT intervention arm will receive the decision aid in addition to enhanced usual care
  Interventions: Other: RECONJOINT
- RCT Participants (Physicians) (Experimental): Participating surgeons will be randomized to Enhanced Usual Care or Intervention with a 1:1 ratio
  Interventions: Other: RECONJOINT

INTERVENTIONS:
Other: RECONJOINT — RECONJOINT is a Breast Reconstruction Decision Aid
  Arms: RCT Participants (Physicians); RECONJOINT/RCT Participants (Patients)

SUMMARY:
The purpose of this study is to find out whether it is practical (feasible) to do a larger study looking at the effectiveness of the Breast Reconstruction Decision Aid Tool (RECONJOINT) for breast reconstruction surgery.

ELIGIBILITY:
Participant Inclusion Criteria

Focus Group Participants

* A diagnosed genetic predisposition to breast cancer or a diagnosis of ductal carcinoma in situ or any invasive cancer confirmed through review of the medical record
* ≥18 years old
* Considering post-mastectomy breast reconstruction

RCT Participants (Patients)

* A diagnosed genetic predisposition to breast cancer or a diagnosis of ductal carcinoma in situ or any invasive cancer confirmed through review of the medical record
* ≥18 years old
* Considering post-mastectomy breast reconstruction
* Have an appointment scheduled for consultation with a plastic surgery provider

RCT Participants (Physicians)

* Provides breast reconstruction care ≥ 50% of the time. This is defined as over half of the surgeon's cases in the preceding calendar year being related to breast reconstruction surgery.

Participant Exclusion Criteria

Focus Group Participants

* Not considering post-mastectomy breast reconstruction
* Non-English proficiency

RCT Participants (Patients)

* Not considering postmastectomy breast reconstruction
* Recurrent or metastatic breast cancer
* Male sex
* Non-English proficiency

RCT Participants (Physicians)

* Does not provide breast reconstruction care at least 50% of the time
* Non-English proficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2029-01-05 (Estimated); Study Completion 2029-01-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility determined by participant accrual | <60 days after initial reconstructive surgery consult and before pt's breast reconstruction surgery
  Determine the feasibility of a hybrid effectiveness-implementation study that investigates the effectiveness and implementation potential of a decision aid to improve shared decision-making in breast reconstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Evan Matros, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Rockville Centre, New York
  - Duke Cancer Institute (Data collection only), Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org